CLINICAL TRIAL: NCT06546956
Title: Developing and Testing a Multicomponent Breathwork Intervention for Adults With Chronic Pain
Brief Title: Integrative Breathwork Intervention for Chronic Pain
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202202844; K01AT012066 (NIH)
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic pain; Breathwork; Mindfulness; Breathing
MeSH Terms: conditions — Chronic Pain; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrative Breathwork Intervention (Experimental): The integrative, multicomponent breathwork intervention that will be tested in this study is called Guided Respiration Mindfulness Therapy. Participants will receive a 60 minute breathwork session once a week for 8 weeks.
  Interventions: Behavioral: Integrative Breathwork Intervention

INTERVENTIONS:
Behavioral: Integrative Breathwork Intervention — GRMT has three core components: respiratory regulation (i.e., sustained conscious connected breathing pattern into the upper chest where there is no pause between inhale and exhale), mindfulness of somatic sensations while breathing (i.e., interoceptive awareness with acceptance), and relaxation of physical tension. These components are the primary focus in every breathwork session. The intervention is delivered 1-on-1 in-person with a trained facilitator. Participants lay supine throughout the 60 minute session. The facilitator observes the participant's breathing pattern and guides the participant to apply the three core components. Each session ends with spontaneous, relaxed breathing and an opportunity to briefly share what happened during the session.
  Other Names: Guided Respiration Mindfulness Therapy (GRMT)

SUMMARY:
The proposed research is to develop and refine a multicomponent breathwork intervention, Guided Respiration Mindfulness Therapy, and to iteratively evaluate its feasibility, acceptability, and plausibility for clinically significant effects in people with chronic low back pain. This integrative breathwork intervention involves a 60-minute breathing session where the focus is to maintain a conscious connected breathing pattern (no pause between inhale and exhale), apply mindful acceptance to somatic sensations, and relax any physical tension. Each breathwork session will be delivered 1-on-1 in person by a trained facilitator. The treatment consists of 8 breathwork sessions, once per week for 8 weeks.

DETAILED DESCRIPTION:
Multiple single-arm iterations of an 8-week breathwork intervention will be conducted to refine and optimize the intervention and protocol. Upon completion of each iteration, quantitative and qualitative data will be gathered to identify possible modifications before proceeding with the next iteration. This work will provide initial evidence on the feasibility, acceptability, and plausibility of clinically significant effects of this type of multicomponent breathwork intervention for adults with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-70 years of age.
* Chronic primary low back pain that has persisted for at least 3 months and on most days for the past 6 months.
* Average pain intensity of ≥ 4/10 for the past month.
* Fluent in English.
* Access to internet with a valid email address.
* Able to lay down and stay relatively still for one hour.

Exclusion Criteria:

* Leg pain, or any other chronic pain, that is greater than low back pain.
* Back pain possibly due to specific conditions (e.g., cancer, infection).
* Ongoing legal action or disability claim related to low back pain.
* Neurological symptoms associated with low back pain, including loss of control or incontinence of bowel or bladder.
* Systemic rheumatic disease/condition (e.g. rheumatoid arthritis, systemic lupus erythematosus, fibromyalgia).
* Respiratory disorder (e.g., chronic obstructive pulmonary disease) or moderate to severe asthma within the past 12 months.
* Activity limiting heart disease including cardiovascular or peripheral arterial disease.
* Uncontrolled hypertension (i.e. SBP/DBP of > 160/95) or orthostatic hypotension (e.g., issues with fainting).
* Neurological disease (e.g. Parkinson's, multiple sclerosis, epilepsy, history of seizures) or evidence of previous brain injury, including stroke and traumatic brain injury.
* Serious acute physical injuries or any surgery within the past 6 months.
* Serious psychiatric disorder (e.g., schizophrenia) or mental health issues requiring hospitalization within the past 12 months or currently on anti-psychotic medications.
* History of hospitalization or treatment of substance use disorder within the past 12 months.
* Currently undergoing curative or palliative chemotherapy or radiation. Pregnant or plan to become pregnant during the study period.
* Glaucoma or detached retina.
* Current participation or participation in the past 2 months of an interventional research study.
* Cognitive impairment or factors that would preclude comprehension of material and/or full participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2027-05-22 (Estimated)

PRIMARY OUTCOMES:
Treatment Acceptability | Post-treatment (after the 8-week intervention)
  Treatment acceptability and participant satisfaction of the breathwork intervention will be measured using the Client Satisfaction Questionnaire and several face valid items. (0-10; higher values = greater treatment acceptability and satisfaction).
Intervention Adherence | Post-treatment (Week 8)
  Percentage of intervention sessions attended by participants.
Participant Retention | Post-treatment (Week 8)
  Percentage of randomized participants who complete post-treatment assessment.
Change in Pain Intensity | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  The Pain, Enjoyment, and General Activities (PEG-3) scale will be used to assess pain intensity over the past week on average. (0-10; higher values = greater pain intensity).
Change in Pain Interference | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  The Pain, Enjoyment, and General Activities (PEG-3) will be used assess pain interference over the past week. (0-10; higher values = greater pain interference).

SECONDARY OUTCOMES:
Treatment Credibility | After Intervention session 3
  Assessed using the 8-item Credibility and Expectancy Questionnaire where higher scores represent higher levels of treatment credibility. (1-9; higher values = greater treatment expectancy and credibility).
Acute Treatment Effects | Before and after each intervention sessions (Weeks 1-8)
  Assessed using face-valid items related to feelings and emotions immediately before and after each intervention session. Change scores will be calculated from post-intervention to pre-intervention. (0-4; higher scores = greater changes in acute subjective effects).
Change in Pain Catastrophizing | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the 13-item Pain Catastrophizing Scale. (Scores range from 0-52; higher scores represent higher levels of pain catastrophizing).
Change in Pain Self-Efficacy | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the 10-item Pain Self-Efficacy Scale. (0-6; higher scores represent higher levels of pain self-efficacy).
Change in Fear Avoidance Beliefs | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the 5-item Fear-Avoidance Beliefs Questionnaire-physical activity subscale. (0-6; higher scores represent higher levels of physical activity-related fear-avoidance beliefs).
Change in Physical Function | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  The PROMIS Physical Function-6b will be used assess pain dysfunction. (1-5; higher scores represent higher levels of physical function).
Change in Sleep Disturbance | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the PROMIS-Sleep Disturbance 8b scale. (1-5; higher scores represent higher levels of sleep disturbance).
Change in Sleep Related Impairment | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the PROMIS-Sleep Related Impairment 8a scale. (1-5; higher scores represent higher levels of sleep related impairment).
Change in Fatigue | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the PROMIS Fatigue-8a scale. (1-5; higher scores represent higher levels of fatigue over the past week).
Change in Stress | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the 4-item Perceived Stress Scale. (0-4; higher scores represent higher levels of subjective stress over the past month).
Change in Anxiety | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the Generalized Anxiety Disorder-2 Questionnaire. (0-3; higher scores represent higher levels of anxiety over the past 2 weeks).
Change in Depression | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the Patient Health Questionnaire-2.(0-3; higher scores represent higher levels of depression over the past 2 weeks).
Change in Multisensory Sensitivity | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the Multisensory Amplification Scale will be used to assess symptoms of central nervous system hypersensitivity, or central sensitization. (1-5; higher scores represent higher levels of sensory sensitivity).
Change in Interoception | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the Multidimensional Assessment of Interoceptive Awareness-2. (0-5; higher scores represent higher levels of interoception).
Change in Mindful Reappraisal of Pain Sensations | Change from Baseline (Week 0) to Post-treatment (Week 8), 1-month follow-up.
  Assessed using the Mindful Reappraisal of Pain Sensations Scale. (0-6; higher scores represent higher levels of mindful reappraisal).

OTHER OUTCOMES:
Psychological Insight | Post-treatment (Week 8)
  Assessed using the Psychological Insight Questionnaire. (0-5; higher scores represent greater levels of psychological insight).

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pratscher, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States